CLINICAL TRIAL: NCT01753349
Title: An International Observational Prospective Study On Long-Term Response To Botulinum Toxin Type A (BoNT-A) Injections In Subjects Suffering From Idiopathic Cervical Dystonia (CD) - Pharmaco-Economic Impact
Brief Title: Phase IV-Cervical Dystonia-INTEREST IN CD2
Acronym: INTEREST_INCD2
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: Y-79-52120-166
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Idiopathic cervical dystonia: Adults subjects from Hospitals, Private Practices suffering idiopathic cervical dystonia. BoNT-A injections, 3-4 times yearly.
  Interventions: Biological: Botulinum toxin type A

INTERVENTIONS:
Biological: Botulinum toxin type A — Investigators were free to prescribe any BoNT A preparation, including Dysport, Botox and Xeomin.

SUMMARY:
The purpose of the study is to document long-term response in real-life practice after injection cycles with BoNT-A in subjects suffering from idiopathic cervical dystonia (Long-term clinical and pharmaco-economic data).

ELIGIBILITY:
Inclusion Criteria:

* Subject for whom there is an intention to treat with BoNT-A.
* BoNT treatment naïve or previously treated with BoNT.
* If previously treated with BoNT, at least a 12-week interval between the last injection (BoNT-A or BoNT-B) and inclusion.
* Subject able to comply with the protocol.
* Provision of written informed consent prior to collect the data.

Exclusion Criteria:

* Contraindications to any BoNT-A preparations.
* The subject has already been included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects from Hospitals, Private Practices suffering idiopathic cervical dystonia.
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09-25 (Actual)

PRIMARY OUTCOMES:
Change in subject's satisfaction using a 5-point Likert scale. | Baseline and at every 3 to 4 months, up to 3 years.
  Identification of prognostic factors for subject's satisfaction regarding control of symptoms associated with idiopathic CD.

SECONDARY OUTCOMES:
Change from baseline in Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) total score and severity sub-scale. | Baseline and at every 3 to 4 months, up to 3 years.
  Assessment of severity of CD.
Change in tremor associated with CD using Tsui score | Baseline and at every 3 to 4 months, up to 3 years.
Change in pain relief assessed using the TWSTRS pain sub-scale. | Baseline and at every 3 to 4 months, up to 3 years.
Change in disability will be measured with the TWSTRS disability sub-scale. | Baseline and at every 3 to 4 months, up to 3 years.
Pharmaco-economic endpoints | Baseline and at every 3 to 4 months, up to 3 years.
  * Time intervals between injections
  * Changes in concomitant treatments for CD and associated symptoms.
  * Changes in employment status

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (113):
- United States (4):
  - Parkinson's and Movement Disorders Center of Maryland, Elkridge, Maryland
  - Tufts Medical Center, Inc, Boston, Massachusetts
  - The Parkinson's and Movement Disorders Center, Southfield, Michigan
  - Vanderbilt University, Nashville, Tennessee
- Algeria (3):
  - Bab El Oued Hospital, Algiers
  - Sidi Bel Abbes Hospital, Algiers
  - Ben Badis Hospital, Constantine
- Australia (5):
  - Austin Hospital, Heidelberg, Victoria
  - Alfred Hospital,, Melbourne
  - Dandenong Neurology, Melbourne
  - Royal North Shore Hospital, Sydney
  - Burwest Neurophysiology, Sydney
- Medical University of Vienna Spitalgasse 23, Vienna, Austria
- Belgium (4):
  - AZ Sint Jan Brugge - Oostende AV, Bruges
  - Universitair Ziekenhuis Antwerpen, Edegem
  - AZ Sint Lucas, Ghent
  - Centre Hospitalier Universitaire de Liège, Liège
- Brazil (4):
  - Hospital das Clínicas, Universidade Federal de Minas Gerais, Belo Horizonte
  - Campus Universitario, Ribeirão Preto
  - Hospital Universitario Antoni Pedro, Rio de Janeiro
  - Instituto de Medicina Física e Reabilitaçao, São Paulo
- Queen Mary Hospital, Hong Kong, China
- Czechia (4):
  - Faculty Hospital Sv. Anna Brno, Brno
  - Faculty hospital Olomouc, Olomouc
  - Pardubice Regional Hospital, Inc., Pardubice
  - Department of Neurology 1st LF UK and VFN, Prague
- Estonia (2):
  - East Tallinn Central Hospital, Tallinn
  - Tartu University Hospital, Neurology Clinic, Tartu
- France (8):
  - Centre Hospitalier d'Albi, Albi
  - CHU Amiens Nord, Amiens
  - CHI Robert Ballanger, Aulnay-sous-Bois
  - CHRU Lyon Est Hôpital Neurologique et Neurochirurgical Pierre Wertheimer, Bron
  - Hôpital Roger Salengro, Lille
  - Hôpital La Timone, Marseille
  - Hopital universitaire Carémeau, Nîmes
  - Hôpital Purpan, Toulouse
- Germany (6):
  - Neurologische Universitätsklinik Erlangen, Erlangen
  - Neurologische Privatpraxis, Hanover
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - Hauptstraße 1a, Neusaß
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Würzburg, Würzburg
- Hungary (2):
  - Semmelweis Egyetem, Budapest
  - Jósa András Oktató Kórház, Nyíregyháza
- Israel (3):
  - Carmel Medical Center Haifa Israël, Haifa
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (8):
  - Ospedali Riuniti di Bergamo, Bergamo
  - Azienda Ospedaliera-Universitaria, Ferrara
  - A.O.U. Policlinico "G. Martino, Messina
  - II Università degli Studi di Napoli, Napoli
  - A.O. Villa Sofia CTO, Palermo
  - Policlinico Umberto I, Università La Sapienza, Roma
  - Università La Sapienza, Roma
  - Ospedale Mauriziano - Umberto I, Torino
- Jordan Hospital, Amman, Jordan
- Latvia (2):
  - National Rehabilitation center "Vaivari", Jūrmala
  - P. Stradins Clinical University hospital, Riga
- Lebanon (2):
  - Hopital Hotel Dieu, Beirut
  - Centre Hospitalier Universitaire Notre Dame de Secours, Byblos
- Malaysia (2):
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University of Malaysia, Kuala Lumpur
- Mexico (6):
  - Centro Medico Zambrano Hellion, San Pedro Garza García, Nuevo León
  - Hospital General Dr. Santiago Ramón y Cajal, Durango
  - Hospital General de México, Mexico City
  - Nuevo Hospital Obregón, Mexico City
  - Instituto Nacional de Neurología y Neurocirugía "Manuel Velasco Suárez", Mexico City
  - Centro de Rehabilitación Integral de Querétaro, Querétaro
- Philippines (2):
  - Metropolitan Medical Center, Manila
  - St Luke's Medical Center, Quezon
- Poland (2):
  - Specjalistyczna Praktyka Lekarska, Katowice
  - Medical University of Warsaw, Warsaw
- Portugal (4):
  - Centro Hospitalar Lisboa Norte, Lisbon
  - Centro Hospitalar do Porto, Porto
  - Hospital São Bernardo, Setùbal
  - Centro Hospitalar de Trás-os-Montes e Alto Douro, Vila Real
- Romania (2):
  - Spitalul Universitar de Urgenta Bucuresti, neurologie, Bucharest
  - Spitalul Clinic Judetean de Urgenta Timisoara, neurologie II, Timișoara
- Russia (5):
  - The Chelyabinsk state medical academy,, Chelyabinsk
  - State Institution "Interregional clinical diagnostic centre", Kazan'
  - State Educational Institution of high professional education "Krasnoyarsk State Medical University named after Professor V.F. Voyno-Yasenetsky of the Ministry of Health and Social Development of Russia", Krasnoyarsk
  - State Federal Budgetary Institution Scientific Center of Neurology RAMS, Moscow
  - State Educational Institution of high professional education "St-Peterbusrg state medical university named after I.P. Pavlov of Roszdrav", St-Peterburg
- Serbia (2):
  - Clinical Center of Serbia, Belgrade
  - Military Medical Academy, Belgrade
- Singapore General Hospital, Singapore, Singapore
- Slovenia (2):
  - University Medical Centre Ljubljana, Ljubljana
  - University Clinical Centre Maribor, Maribor
- South Korea (5):
  - Dong-A University Hospital, Busan
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Sweden (6):
  - Stortorgets Neurologmottagning, Helsingborg
  - Universtitessjukhuset i Linköping, Linköping
  - Skånes University Hospital, Malmo
  - Neuroenheten Utsikten, Stockholm
  - Norrlands Universitetssjukhus (NUS), Umeå
  - Uppsala University Hospital, Uppsala
- Taiwan (3):
  - Kaohsiung Chang-gung Memorial Hospital, Kaohsiung City
  - TaiChung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Thailand (2):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Siriraj Hospital, Bangkok
- Turkey (Türkiye) (4):
  - Gazi University Medical Faculty, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Istanbul University Cerrahpaşa Medical Faculty, Istanbul
  - Dogu Mersin University Hospital, Mersin
- Rashid Hospital, Dubai, United Arab Emirates
- United Kingdom (4):
  - Royal Devon & Exeter Hospital, Exeter
  - Leeds General Infirmary, Leeds
  - Neurology, John Radcliffe Hospital, Oxford
  - Queen's Hospital Romford, Romford

REFERENCES:
- [Derived] Trosch RM, Misra VP, Maisonobe P, Om S. Impact of abobotulinumtoxinA on the clinical features of cervical dystonia in routine practice. Clin Park Relat Disord. 2020 Jun 15;3:100063. doi: 10.1016/j.prdoa.2020.100063. eCollection 2020. PMID 34316644